CLINICAL TRIAL: NCT00825734
Title: Phase I/II Trial of Sorafenib Plus Ixabepilone in HER2-Negative Metastatic Breast Cancer (MBC)
Brief Title: Phase I/II Trial of Sorafenib Plus Ixabepilone in HER2-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bayer (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 138
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Sorafenib; Nexavar; Ixabepilone; Ixempra
MeSH Terms: conditions — Breast Neoplasms | interventions — Sorafenib; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Level 1 (Experimental): Sorafenib PO BID (200mg), Ixabepilone IV every 21 days (40mg/m^2)
  Interventions: Drug: Sorafenib; Drug: Ixabepilone
- Dose Level -1 (Experimental): Sorafenib PO BID (200mg), Ixabepilone IV every 21 days (32mg/m^2)
  Interventions: Drug: Sorafenib; Drug: Ixabepilone
- Dose Level 1a (Experimental): Sorafenib PO BID (400mg), Ixabepilone IV every 21 days (32mg/m^2)
  Interventions: Drug: Sorafenib; Drug: Ixabepilone

INTERVENTIONS:
Drug: Sorafenib — Dose Level 1 - Sorafenib PO BID (200mg) Dose Level -1 - Sorafenib PO BID (200mg) Dose Level 1a - Sorafenib PO BID (400mg)
  Other Names: Nexavar (Sorafenib)
Drug: Ixabepilone — Dose Level 1 - Ixabepilone IV every 21 days (40mg/m^2) Dose Level -1 - Ixabepilone IV every 21 days (32mg/m^2) Dose Level 1a - Ixabepilone IV every 21 days (32mg/m^2)
  Other Names: Ixempra (Ixabepilone)

SUMMARY:
In this study, patients with metastatic HER2-negative breast cancer will receive treatment with ixabepilone and sorafenib until disease progression or unacceptable toxicity occurs. The Phase I portion of this study will determine the maximum tolerated doses (MTDs) of sorafenib and ixabepilone that may be used in combination for first- or second-line treatment of MBC. The MTDs identified in the Phase I portion of the study will be used in the Phase II portion which will evaluate the efficacy and safety of the combination of sorafenib and ixabepilone in patients who have received at least one prior chemotherapy treatment in either the adjuvant or neoadjuvant setting or following one prior MBC chemotherapy in MBC patients who had not received prior adjuvant or neoadjuvant breast cancer chemotherapy. This will be one of the initial trials investigating the use of this treatment combination for MBC.

This trial will be conducted under the leadership of the Sarah Cannon Research Institute (SCRI) Oncology Research Consortium, a community-based, multi-center, clinical trial organization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically or cytologically confirmed breast cancer diagnosis

with metastatic disease. Patients without pathologic or cytologic

confirmation of metastatic disease should have unequivocal

evidence of metastasis.

3. Measurable disease, as per RECIST criteria (Therasse et al.

2000). Measurable disease cannot be previously irradiated

unless progression was documented. Measurable disease is

defined as: at least one lesion that can be accurately measured in

at least one dimension [longest diameter to be recorded] as

>20 mm with conventional techniques, or as >10 mm with spiral

computed tomography (CT) scan. Disease must be measurable,

i.e., bone-only disease or evaluable-only disease is not eligible.

4. Patients with brain metastasis may participate if they:

• have undergone appropriate treatment,

* are at least 1 month post-treatment,
* have no neurologic symptoms,
* are not on steroids,
* have a follow-up magnetic resonance imaging (MRI) scan that

demonstrates no residual active lesions, and

* have no new untreated lesions.

  5 The following prior therapies are allowed:
* No prior chemotherapy in the metastatic setting. However,

patients must have received prior adjuvant or neo-adjuvant

chemotherapy.

* Prior radiation therapy in either the metastatic or early-stage

setting, as long as <25% of the bone marrow has been

treated. Radiation therapy must be completed at least

14 days prior to study registration, and all radiation-related

toxicities must be resolved to ≤ grade 1 before the patient is

eligible for study inclusion.

* Any number of hormonal therapies in the neo-adjuvant,

adjuvant, or metastatic setting is allowed. Patients must

discontinue hormonal therapy at least 1 week prior to starting

study treatment.

•Prior bevacizumab administered >4 weeks before initiation of

study treatment is allowed.

6 HER2-negative status. Documentation of HER2 results must be

available at the time of study enrollment. HER2-negative is

defined as:

* Immunohistochemical (IHC) 0 or IHC 1+ OR
* Fluorescence in situ hybridization (FISH) negative (defined by

FISH ratio <2.2) OR

* Silver in-situ hybridization (SISH) negative (defined by SISH

ratio <2.2).

Patients with an IHC 2+ will need to be validated as HER2-negative

by FISH.

7 An Eastern Cooperative Oncology Group (ECOG) performance

status of < or = to 2.

8. Normal bone marrow function as defined by:

* absolute neutrophil count (ANC) >1,500/μL;
* platelets >100,000/μL;
* hemoglobin >9 g/dL.

  9 Normal hepatic function as defined by:
* total bilirubin within normal institutional limits;
* aspartate aminotransferase (AST) and alanine

aminotransferase (ALT) <2.5 × the institutional upper limit of

normal (ULN) for patients without liver metastasis; <5.0 × ULN

for patients with liver metastasis.

10. Normal renal function as defined by creatinine <1.5 × ULN.

11. Left ventricular ejection fraction (LVEF) within institutional limits of

normal.

12. International normalized ratio (INR) <1.5 or a prothrombin

time/partial thromboplastin time (PT/PTT) within normal limits.

Patients receiving anti-coagulation treatment with an agent such

as warfarin or heparin may be allowed to participate. The INR

should be measured prior to initiation of sorafenib, and for

patients on warfarin, INR should be monitored at least weekly

following initiation of protocol treatment, until the INR is stable and

therapeutic.

13. Life expectancy of >6 months.

14. For women of childbearing potential, negative serum pregnancy

test within 7 days prior to starting treatment.

15. For women of childbearing potential and men, agreement to use a

method of contraception that is acceptable to their physician from

time of first signing the informed consent and for the study

duration. Men should use adequate birth control for at least three

months after the last administration of sorafenib. If a woman

becomes pregnant or suspects she is pregnant while participating

in this study, she must agree to inform her treating physician

immediately. As applicable, patients must agree to discontinue

breast-feeding until at least 3 weeks after their last dose of study

drug.

16. Recovery to < grade 1 toxicity due to prior therapy.

17. Ability to understand and willingness to sign a written informed

consent document.

Exclusion Criteria

1. More than one (>1) prior chemotherapy regimen.
2. Treatment with chemotherapy, biologic agents, or targeted agents

   within the previous 4 weeks.
3. Previous treatment with sorafenib or ixabepilone.
4. Women who are pregnant or breastfeeding.
5. Neuropathy (motor or sensory) greater than grade 1.
6. Uncontrolled intercurrent illness including (but not limited to)

   ongoing or active infection >grade 2.
7. Known history of human immunodeficiency virus (HIV), Hepatitis

   B, or Hepatitis C infection.
8. History of other non-breast cancer malignancy treated with

   curative intent within the 5 years preceding study enrollment with

   the exception of carcinoma in situ of the cervix, non-melanoma

   skin cancer, or follicular thyroid cancer.
9. Concurrent hormonal therapy, chemotherapy other than

   ixabepilone, or radiation treatments while on study as well as

   treatment with other investigational agents while on study.
10. Cardiac disease:

    •Congestive heart failure (CHF) greater than New York Heart Association

    (NYHA) Class II (see Appendix B).
    * Unstable angina (anginal symptoms at rest) or new onset angina

      (i.e., began within the last 3 months).
    * Myocardial infarction within the past 6 months.
    * Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
11. Uncontrolled hypertension (systolic blood pressure >150 mmHg

    or diastolic pressure >100 mmHg despite optimal medical

    management).
12. Thrombolic or embolic events such as cerebrovascular accident,

    including transient ischemic attacks, within the past 6 months.
13. Pulmonary hemorrhage or bleeding event ≥ grade 2 within

4 weeks of the first dose of study treatment, or any other

hemorrhage or bleeding event ≥ grade 3 within 4 weeks of the

first dose of study treatment.

14. Serious non-healing wound, ulcer, or bone fracture.

15. Evidence or history of bleeding diathesis or coagulopathy.

16. Major surgery, open biopsy or significant traumatic injury within

4 weeks of the first dose of study drugs or anticipation of the need

for major surgical procedure.

17. Chronic use of CYP3A4 inducers and use of the following strong

CYP3A4 inhibitors: ketoconazole, itraconazole, clarithromycin,

atazanavir, nefazodone, saquinavir, telithromycin, ritonavir,

amprenavir, indinavir, nelfinavir, delavirdine, and voriconazole.

Use of these agents should be discontinued at least 72 hours

prior to initiation of study treatment.

18. Use of St. John's Wort or rifampin (rifampicin).

19. Any condition that impairs patient's ability to swallow whole pills or

gastrointestinal (GI) tract disease that involves an inability to take

oral medication, malabsorption syndrome, a requirement for

intravenous (IV) alimentation, prior surgical procedures affecting

absorption, or uncontrolled inflammatory GI disease (e.g., Crohn's

disease or ulcerative colitis).

20. Psychiatric illness/social situations that would limit compliance

with study requirements.

21. Known or suspected allergy to sorafenib, Cremophor EL

(polyoxyethylated castor oil) or a drug formulated in

Cremophor EL such as paclitaxel or any other agent given in the

course of this trial.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-03; Primary Completion 2013-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (15):
- United States (15):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Providence Medical Group, Terre Haute, Indiana
  - RHHP/ Hope Cancer Center, Terre Haute, Indiana
  - Baptist Hospital East, Louisville, Kentucky
  - Hematology Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Mercy Hospital, Portland, Maine
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at multiple dose levels into the Dose Escalation (Phase I) portion of this study to determine the safest dose of this regimen (MTD-Maximum Tolerated Dose). Upon determination of this dose, patients being treated at the MTD proceeded to the Dose Expansion (Phase II) portion of the study and additional patients were recruited
Period: Phase I
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level 1a
Started | 4 | 3 | 3
Completed | 0 (Patients were on-study until determination of the Maximum Tolerated Dose (MTD)) | 0 (Patients were on-study until determination of the Maximum Tolerated Dose (MTD)) | 3
Not Completed | 4 | 3 | 0
Period: Phase II
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level 1a
Started | 0 | 0 | 76 (Includes patients treated at MTD during Phase I and 73 additional patients enrolled for Phase II)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 76

BASELINE CHARACTERISTICS:
Groups:
- All Patients: Patients treated at all dose levels in the Phase I and Phase II portions of the study
  : Dose Level 1 (4 patients) Sorafenib PO BID (200mg), Ixabepilone IV every 21 days (40mg/m^2)
  Dose Level -1 (3 patients) Sorafenib PO BID (200mg), Ixabepilone IV every 21 days (32mg/m^2)
  Dose Level 1a (76 patients) Sorafenib PO BID (400mg), Ixabepilone IV every 21 days (32mg/m^2)
Arm/Group | All Patients
Number analyzed (Participants) | 83
Age, Continuous [Median (Full Range); unit: Years] | 57 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 83

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Measured from Day 1 of study drug administration to disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) - progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: every 9 weeks until treatment discontinuation or death on study
Population: Includes patients treated at the Phase II dose
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Sorafenib and Ixabepilone: Oral targeted therapy and Systemic Chemotherapy
Arm/Group | Sorafenib and Ixabepilone
Number analyzed (Participants) | 76
months | 4.8 [3.5 to 6.3]

2. Secondary Outcome: 6-month Progression-Free Survival
Description: Measured from Day 1 of study drug administration to disease progression as defined by RECIST v1.1, or death on study. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: every 9 weeks, up to 6 months
Population: Includes patients treated at the Phase II dose
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib and Ixabepilone
Number analyzed (Participants) | 76
percentage of participants | 42

3. Secondary Outcome: Objective Response Rate
Description: Objective Response will be evaluated in this study using the Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: every 9 weeks until discontinuation of treatment
Population: Includes patients treated at the Phase II dose who were evaluable for response
Measure: Number; unit: patients
Arm/Group | Sorafenib and Ixabepilone
Number analyzed (Participants) | 68
patients | 28

4. Secondary Outcome: Overall Survival (OS)
Description: Measured from Day 1 of study drug administration to date of death due to any cause.
Time Frame: every 9 weeks until treatment discontinuation or death on study
Population: Includes patients treated at the Phase II dose
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib and Ixabepilone
Number analyzed (Participants) | 76
months | 15.5 [11 to 20.6]

5. Secondary Outcome: Number of Patients With Adverse Events as a Measure of of Safety and Tolerability
Description: Assessments are made through analysis of reported incidence of treatment-emergent AEs and SAEs.
Time Frame: every 9 weeks until treatment discontinuation or unacceptable toxicity
Population: Patients treated at the Phase II dose
Measure: Number; unit: participants
Groups:
- Phase II - Sorafenib and Ixabepilone: Oral targeted therapy and Systemic Chemotherapy
Arm/Group | Phase II - Sorafenib and Ixabepilone
Number analyzed (Participants) | 76
participants
  Neutropenia | 33
  Febrile neutropenia | 1
  Anemia | 27
  Thrombocytopenia | 22
  Fatigue | 54
  Nausea/vomiting | 54
  Rash | 40
  Neuropathy | 39
  Anorexia/weight loss | 36
  Diarrhea | 33
  Arthralgia/myalgia | 32
  Alopecia | 30
  Pain in extremity | 18
  Hypertension | 18
  Constipation | 17
  Dyspnea | 12
  Hand-foot syndrome | 12
  Taste alteration | 11
  Mucositis | 10
  Pruritus | 9

ADVERSE EVENTS:
Groups:
- Dose Level 1a: Includes patients treated at the Phase II dose - Sorafenib PO BID (400mg), Ixabepilone IV every 21 days (32mg/m^2)
Arm/Group | Dose Level 1a
Serious Adverse Events (participants affected / at risk) | 6/76
Other Adverse Events (participants affected / at risk) | 75/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1a (N=76)
ACUTE RENAL FAILURE (Renal and urinary disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (3)
DEATH (General disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
INFECTION (Infections and infestations) | 1 (2)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
WEIGHT LOSS (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1a (N=76)
ABDOMINAL PAIN (Gastrointestinal disorders) | 10 (41)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 4 (16)
ALLERGIC REACTION (Immune system disorders) | 10 (11)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 7 (26)
ALOPECIA (Skin and subcutaneous tissue disorders) | 31 (174)
ANEMIA (Blood and lymphatic system disorders) | 27 (119)
ANOREXIA (Metabolism and nutrition disorders) | 28 (76)
ANXIETY (Psychiatric disorders) | 6 (23)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 29 (106)
ASTHENIA (Musculoskeletal and connective tissue disorders) | 14 (99)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 (49)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 8 (19)
CALLUS (Skin and subcutaneous tissue disorders) | 5 (41)
CHEST PAIN (General disorders) | 14 (26)
CHILLS (General disorders) | 4 (7)
CONSTIPATION (Gastrointestinal disorders) | 24 (56)
COUGH (Respiratory, thoracic and mediastinal disorders) | 19 (55)
DEHYDRATION (Metabolism and nutrition disorders) | 6 (7)
DEPRESSION (Psychiatric disorders) | 7 (31)
DESQUAMATION (Skin and subcutaneous tissue disorders) | 6 (11)
DIARRHEA (Gastrointestinal disorders) | 35 (126)
DIZZINESS (Nervous system disorders) | 12 (43)
DRY MOUTH (Gastrointestinal disorders) | 4 (17)
DRY SKIN (Skin and subcutaneous tissue disorders) | 9 (58)
DYSPEPSIA (Gastrointestinal disorders) | 8 (35)
DYSPHAGIA (Gastrointestinal disorders) | 4 (4)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 23 (79)
EDEMA (General disorders) | 15 (36)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 6 (10)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5 (11)
FATIGUE (General disorders) | 61 (274)
FEVER (General disorders) | 10 (19)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 5 (7)
FLUSHING (Vascular disorders) | 4 (10)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 (17)
HEADACHE (Nervous system disorders) | 13 (29)
HOT FLASHES (Vascular disorders) | 4 (18)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 8 (31)
HYPERTENSION (Vascular disorders) | 26 (104)
HYPOKALEMIA (Metabolism and nutrition disorders) | 5 (21)
HYPOTENSION (Vascular disorders) | 5 (5)
INFECTION (Infections and infestations) | 9 (10)
INSOMNIA (Psychiatric disorders) | 11 (63)
LEUKOPENIA (Blood and lymphatic system disorders) | 32 (114)
LYMPHEDEMA (Vascular disorders) | 4 (8)
MUCOSITIS (Gastrointestinal disorders) | 13 (23)
MYALGIA (Musculoskeletal and connective tissue disorders) | 15 (42)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 5 (12)
NASAL DRAINAGE (Respiratory, thoracic and mediastinal disorders) | 4 (8)
NAUSEA (Gastrointestinal disorders) | 39 (141)
NEUTROPENIA (Blood and lymphatic system disorders) | 36 (115)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 23 (88)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 12 (46)
PERIPHERAL NEUROPATHY (Nervous system disorders) | 41 (255)
PRURITUS (Skin and subcutaneous tissue disorders) | 10 (21)
Pain (General disorders) | 7 (16)
RASH (Skin and subcutaneous tissue disorders) | 41 (158)
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 5 (11)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 6 (11)
TACHYCARDIA (Cardiac disorders) | 6 (19)
TASTE ALTERATION (Nervous system disorders) | 10 (50)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 23 (65)
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 5 (7)
VOMITING (Gastrointestinal disorders) | 20 (37)
WEIGHT LOSS (Investigations) | 11 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other